CLINICAL TRIAL: NCT03365895
Title: Evaluating the Role of Diffusion Tensor Imaging in Predicting Development of Chemotherapy Induced Peripheral Neuropathy in Patients With Breast Cancer
Brief Title: Diffusion Tensor Imaging in Predicting Development of Chemotherapy Induced Peripheral Neuropathy in Patients With Breast Cancer (CIPN)
Acronym: CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1707634514; NCI-2017-01413 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CIPN; 1707634514 (Other: University of Arizona); P30CA023074 (NIH)
Record Dates: First submitted 2017-11-16; First posted 2017-12-07 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Breast Carcinoma; Breast Cancer; Neuropathy;Peripheral; Neuropathy
Keywords: diffusion; tensor; imaging; chemotherapy; peripheral neuropathy; breast cancer; MRI; Magnetic Resonance Imaging; Diffusion Tensor Imaging
MeSH Terms: conditions — Breast Neoplasms; Neuritis; Peripheral Nervous System Diseases | interventions — Diffusion Tensor Imaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (non-enhanced MRI using MRN and DTI) (Experimental): Patients undergo non-enhanced MRI of both lower extremities using MRN and DTI prior to initiation and after completion of standard of care chemotherapy.
  Interventions: Procedure: Diffusion Tensor Imaging; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Diffusion Tensor Imaging — Undergo non-enhanced MRI using MRN and DTI
  Other Names: DIFFUSION TENSOR MRI; DT-MRI; DTI
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo non-enhanced MRI using MRN and DTI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot early phase I trial studies how well diffusion tensor imaging works in predicting development of chemotherapy induced peripheral neuropathy in patients with breast cancer. Diffusion tensor imaging may help to get better pictures of the nerves of feet and lower legs before and after chemotherapy treatment and may help to predict the risk of developing peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the changes in the fractional anisotropy (FA) and apparent diffusion coefficient (ADC) values of the lower extremity nerves by diffusion tensor imaging (DTI) before initiation and after completion of taxane chemotherapy in patients with breast cancer.

SECONDARY OBJECTIVES:

I. Establish normal and abnormal FA and ADC values of the lower extremity nerves.

II. Evaluate relationship of DTI findings of chemotherapy induced peripheral neuropathy (CIPN) with self-reported Patient Neurotoxicity Questionnaire (PNQ) and Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-neurotoxicity questionnaire (FACT-GOT-NTX) questionnaires.

III. Assess inter-reader variability in measuring FA and ADC values.

OUTLINE:

Patients undergo non-enhanced magnetic resonance imaging (MRI) of both lower extremities using magnetic resonance neurography (MRN) and DTI prior to initiation and after completion of standard of care chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Be capable of understanding the investigational nature of the study and all pertinent aspects of the study
* Be capable of signing and providing written consent in accordance with institutional and federal guidelines
* Have a histologically-confirmed diagnosis of breast cancer
* Need to be treated with taxane containing chemotherapy as determined by their treating physician
* Be able to undergo magnetic resonance (MR) imaging
* Be willing and able to comply with scheduled visits, treatment plan, and MR imaging

Exclusion Criteria:

* Have non-MRI compatible metallic objects on/in body
* Have metallic hardware in the lower extremity which is MR compatible however would create too much artifact for MR examination
* Are unable to lay still in the MR scanner for length of examination
* Have severe claustrophobia
* Have pre-existing peripheral neuropathy from other medical conditions or due to cancer
* Have diagnosis of diabetes
* Pregnant patients
* Prior exposure to neurotoxic chemotherapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Changes in quantitative fractional anisotropy (FA) of the lower extremity nerves by diffusion tensor imaging (DTI) | Pre-Treatment (0-30 days prior to receiving first chemotherapy) and Post-Treatment (0-30 days after last day of chemotherapy)
  The quantitative DTI parameters measured before the initiation of and after completion of chemotherapy will be compared and used to calculate the degree of change. Descriptive statistics (with confidence interval [CI]) will be used for the current sample size.
Changes in apparent diffusion coefficient (ADC) of the lower extremity nerves by diffusion tensor imaging (DTI) | Pre-Treatment (0-30 days prior to receiving first chemotherapy) and Post-Treatment (0-30 days after last day of chemotherapy)
  The quantitative DTI parameters measured before the initiation of and after completion of chemotherapy will be compared and used to calculate the degree of change. Descriptive statistics (with confidence interval [CI]) will be used for the current sample size.

SECONDARY OUTCOMES:
Inter-reader variability and reproducibility in measuring fractional anisotropy (FA) by diffusion tensor imaging (DTI) | Pre-Treatment (0-30 days prior to receiving first chemotherapy) and Post-Treatment (0-30 days after last day of chemotherapy)
  Inter-reader agreement in measuring the quantitative DTI measurements will be assessed by percentage agreement.
Inter-reader variability and reproducibility in measuring apparent diffusion coefficient (ADC) by diffusion tensor imaging (DTI) | Pre-Treatment (0-30 days prior to receiving first chemotherapy) and Post-Treatment (0-30 days after last day of chemotherapy)
  Inter-reader agreement in measuring the quantitative DTI measurements will be assessed by percentage agreement.
Normal fractional anisotropy (FA) values of lower extremity nerves | Pre-Treatment (0-30 days prior to receiving first chemotherapy) and Post-Treatment (0-30 days after last day of chemotherapy)
  The normal FA and ADC values of the lower extremity nerves will be estimated using mean FA and ADC values with 95% CIs for before and after chemotherapy will be calculated.
Normal apparent diffusion coefficient (ADC) values of lower extremity nerves | Pre-Treatment (0-30 days prior to receiving first chemotherapy) and Post-Treatment (0-30 days after last day of chemotherapy)
  The normal FA and ADC values of the lower extremity nerves will be estimated using mean FA and ADC values with 95% CIs for before and after chemotherapy will be calculated.
Peripheral neuropathy severity questionnaires | Pre-Treatment (0-30 days prior to receiving first chemotherapy) and on last day of chemotherapy
  The correlation between FA and ADC values with the self-reported Patient Neurotoxicity Questionnaire and Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-neurotoxicity questionnaire will be evaluated using Pearson or spearman correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, MPH, Principal Investigator — The University of Arizona Cancer Center; Lana Gimber, MD, MPH, Principal Investigator — The University of Arizona Cancer Center
Locations (1):
- The University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided